CLINICAL TRIAL: NCT03489525
Title: A Phase 1, Open-label Study to Evaluate the Safety, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of MEDI2228 in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: MEDI2228 in Subjects With Relapsed/Refractory Multiple Myeloma
Acronym: MEDI2228
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7900C00001
Record Dates: First submitted 2018-03-17; First posted 2018-04-05 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: multiple myeloma; relapsed/refractory; open-label
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — arginine decarboxylase; Immunoconjugates

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation, MEDI2228, ADC (Experimental): Single agent MEDI2228, ADC (antibody drug conjugate) will be administered to adult subjects with relapsed/refractory (R/R) multiple myeloma (MM).
  Interventions: Biological: Dose Escalation, MEDI2228, ADC (antibody drug conjugate)
- Dose Expansion, MEDI2228, ADC (Experimental): Single agent MEDI2228, ADC (antibody drug conjugate) will be administered to adult subjects with R/R MM in the dose-expansion cohort at the dose selected for evaluation in the dose-expansion phase.
  Interventions: Biological: Dose Expansion, MEDI2228, ADC (antibody drug conjugate)

INTERVENTIONS:
Biological: Dose Escalation, MEDI2228, ADC (antibody drug conjugate) — Single agent MEDI2228 will be administered to adult subjects with R/R MM. The study aims to evaluate up to 9 planned, sequentially ascending main dose levels
  Arms: Dose Escalation, MEDI2228, ADC
Biological: Dose Expansion, MEDI2228, ADC (antibody drug conjugate) — Adult subjects with R/R MM with measurable disease will be enrolled in the dose-expansion cohort at the dose selected for evaluation in the dose-expansion phase.
  Arms: Dose Expansion, MEDI2228, ADC

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and tolerability, describe the dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) or maximum administered dose (MAD [in the absence of establishing the MTD]) for single agent MEDI2228 in adult subjects with multiple myeloma who are either transplant ineligible or post autologous stem cell transplant and are relapsed/refractory.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥ 18 years of age at the time of screening.
2. Subjects must have a confirmed diagnosis of relapsed/refractory MM as per IMWG criteria (Rajkumar et al, 2014) and have exhausted standard of care regimens with proven clinical benefit, which include agents from the following anti myeloma therapies: PIs, IMIDs, and mAbs and have measurable disease with at least one of the following criteria:

   1. Serum M-protein ≥ 0.5 g/dL
   2. Urine M-protein ≥ 200 mg/24 hours
   3. Serum free light chain (FLC) assay: involved FLC level ≥ 10 mg/dL provided serum FLC ratio is abnormal.
3. Subjects must either be ineligible for or post-autologous stem cell transplant.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Adequate organ and marrow functions as determined per protocol-defined criteria.

Exclusion Criteria

Any of the following would exclude the subject from participation in the study:

Target Disease:

1. Subjects who have previously received an autologous stem cell transplant if less than 90 days have elapsed from the time of transplant or the subject has not recovered from transplant associated toxicities prior to the first scheduled dose of MEDI2228
2. Subjects who have previously received an allogeneic stem cell transplant
3. Central nervous system (CNS) involvement(including meningeal involvement) by MRI or cerebrospinal fluid exam
4. Known history of polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes (POEMS) syndrome, plasma cell leukemia, Waldenstrom's macroglobulinemia, or amyloidosis

   Medical History and Concurrent Diseases:
5. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | From time of informed consent through 90 days post end of treatment
  To assess by the occurrence of adverse events (AEs)
Occurrence of SAE (serious adverse events) | From time of informed consent through 90 days post end of treatment
  To assess the occurrence of serious adverse events (SAEs)
Occurrence of DLTs (dose limiting toxicities) | From time of informed consent through 90 days post end of treatment
  To assess by the occurrence of hematologic and non-hematologic toxicities, AEs, and abnormal laboratory results
Number of patients with changes in laboratory parameters from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess serum chemistry, hematology, coagulation and urninalysis
Number of patients with changes in vital signs from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess body temperature, blood pressure and heart rate
Number of patients with changes in elctrocardiogram (ECG) results from baseline | From time of informed consent and up to 21 days post end of treatment
  To assess using 12 lead ECG recordings

SECONDARY OUTCOMES:
MEDI2228 maximum observed concentration for PK | From time of informed consent through 60 days post end of treatment
  To assess the pharmacokinetics of MEDI2228
MEDI2228 area under the concentration-time curve for PK | From time of informed consent through 60 days post end of treatment
  To assess the pharmacokinetics of MEDI2228
MEDI2228 clearance for PK | From time of informed consent through 60 days post end of treatment
  To assess the pharmacokinetics of Medi2228
MEDI2228 terminal half-life for PK | From time of informed consent through 60 days post end of treatment
  To assess the pharmacokinetics of MEDI2228
Number of subjects who develop anti-drug antibodies (ADAs) | From time of informed consents through 60 days post end of treatment
  To assess immunogenicity of MEDI2228
Objective response rate (ORR) | From time of informed consent and up to three years after final patient is enrolled
  To assess the anti-tumor activity of MEDI2228
Clinical benefit rate | From time of informed consent up to three years after final patient is enrolled
  To assess clinical benefit of MEDI2228
Duration of response (DoR) | From time of informed consent and up to three years after final patient is enrolled
  To assess the anti-tumor activity of MEDI2228
Progression free survival (PFS) | From time of informed consent and up to three years after final patient is enrolled
  To assess the anti-tumor activity of MEDI2228
Overall Survival (OS) | From time of informed consent and up to three years after final patient is enrolled
  To assess the anti-tumor activity of MEDI2228

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune LLC, Study Director — Sponsor GmbH
Locations (10):
- United States (7):
  - Research Site, Phoenix, Arizona
  - Research Site, Jacksonville, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Charlotte, North Carolina
  - Research Site, Fairfax, Virginia
- Research Site, Melbourne, Australia
- Research Site, Athens, Greece
- Research Site, Badalona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca/MedImmune group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca/MedImmune will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca/MedImmune will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.